CLINICAL TRIAL: NCT04769336
Title: Effectiveness of Point of Care Complete Blood Cell Count Analyzer in Reducing Time to Results
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Northwestern Medicine (Other)
Responsible Party: Principal Investigator, Andrew Gostine, MD, Anesthesiologist, Northwestern Medicine
Other Study IDs: 21-009-LFH
Record Dates: First submitted 2021-02-21; First posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Laboratory Problem

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patient: Each patient will undergo simultaneous testing with two different CBC analyzers.
  Interventions: Device: Central Lab based CBC; Device: Point of Care CBC

INTERVENTIONS:
Device: Central Lab based CBC — lab samples will be sent to the central lab for CBC analysis
Device: Point of Care CBC — lab samples will be analyzed at point of care

SUMMARY:
The current process for getting complete blood cell counts (CBC) results in the operating room during surgery relies on sending blood samples from the operating room to the hospital's central lab. This workflow is complex and often results in handing off the blood sample to 4 or more different staff members before arriving in the lab for analysis. This often causes delayed CBC results, which may lead to inappropriate or delayed clinical decision making. By providing prompt access to CBC results with the use of a point of care CBC analyzer, the clinical workflow efficiency can be significantly improved. This should resulting in better clinical decision making, reductions in costs, increase in patient satisfaction and facilitation of hospital processes.

ELIGIBILITY:
Inclusion Criteria:

* All English speaking patients, 18 years or older, having surgery in the Lake Forest Hospital operating rooms, with a pre-existing indication for CBC analysis.

Exclusion Criteria:

* All patients not meeting inclusion criteria or protected patient populations, specifically, pregnant women, prisoners, cognitively impaired patients, patients unable to consent, students, employees, and children)

Ages: 10 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients coming for surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Time to result | Through study completion, an average of 1 year
  Time between blood draw and CBC result displayed in Electronic medical record

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Lake Forest Hospital, Lake Forest, Illinois, United States

IPD SHARING:
Plan to Share IPD: No